CLINICAL TRIAL: NCT03497806
Title: PRISM-EXT: An Open-Label Extension of CP101 Trials Evaluating Oral Full-Spectrum Microbiota™ (CP101) in Subjects With Recurrence of Clostridium Difficile Infection
Brief Title: Open-Label Extension of CP101 Trials Evaluating Oral Full-Spectrum Microbiota™ (CP101) in Subjects With Recurrence of Clostridium Difficile Infection
Acronym: PRISM-EXT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Finch Research and Development LLC. (Industry)
Collaborators: Medpace, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP101-CDI-E02
Record Dates: First submitted 2018-04-06; First posted 2018-04-13 (Actual); Results first posted 2022-08-30 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: Clostridium Difficile Infection; Recurrent Clostridium Difficile Infection; C. Diff; CDI; Recurrent C. Diff; rCDI; C. Difficile; Recurrent CDI; FMT; Fecal Microbiota; Fecal Transplant
Keywords: Clostridium Difficile Infection; CP101; Crestovo; FMT; CDI; C. difficile; C. diff; Recurrent Clostridium Difficile Infection; Recurrent C. diff; Recurrent CDI; Finch; Fecal transplant; Fecal microbiota transplant; rCDI; Finch Therapeutics
MeSH Terms: conditions — Clostridium Infections; Diabetes Insipidus, Neurogenic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- High Dose CP101 (Experimental): The active ingredient of CP101, Full-Spectrum Microbiota™, is derived from the stools of normal healthy donors who are highly screened, tested, and monitored in a clinically structured donation program.
  Interventions: Biological: CP101

INTERVENTIONS:
Biological: CP101 — Study drug will be administered at Treatment (Day 1) as an oral dose after cessation of standard-of-care CDI antibiotic treatment of the current episode of recurrent CDI.
  Other Names: Full-Spectrum Microbiota™

SUMMARY:
This is an open-label study evaluating the safety and efficacy of CP101 treatment in 1) Subjects in CDI-001 who had a CDI recurrence within 8 weeks of receiving CP101 or placebo; OR 2) adults with recurrent CDI who are eligible for direct study entry into CP101-CDI-E02. Subjects who are experiencing recurrent CDI will undergo screening procedures. Subjects who meet eligibility criteria will be eligible to be enrolled in he study and administered CP101.

Approximately 200 subjects will receive CP101. The treatment duration will be 1 day. Subjects will be monitored for recurrence of CDI, safety, and tolerability for 24 weeks following receipt of CP101. The primary efficacy and safety endpoints will be evaluated at 8 weeks post treatment, and all subjects will continue to be followed for an additional 16 weeks for safety and recurrence of CDI.

ELIGIBILITY:
1. Ability to provide written informed consent;
2. Previously enrolled in PRISM 3, had a CDI recurrence within 8 weeks of receiving CP101 or placebo, and have completed their PRISM 3 end of study visit; OR recurrent CDI
3. An outpatient prior to Treatment
4. Has received a course of standard-of-care CDI antibiotics for the most recent CDI episode, has had an adequate clinical response, and has completed a washout period.

Exclusion Criteria:

1. Pregnant, breast-feeding, or considering becoming pregnant during the study
2. Prior history, evidence, or diagnosis of inflammatory bowel disease (e.g., Crohn's disease and ulcerative colitis)
3. Any prior diagnosis of diarrhea-predominant irritable bowel syndrome
4. Systemic chemotherapy or radiation for the treatment of cancer during the 60 days prior to consent or planned during the 8 weeks following Randomization
5. Prior fecal transplant for any condition, regardless of route of administration in the last year or plans to undergo during the study
6. Major intra-abdominal surgery within the past 60 days prior to Screening
7. Admitted to, or expected to be admitted to an intensive care unit for any medical reason. Note: Residents of long term care facilities are eligible study entry
8. History of total colectomy/ileostomy or bariatric surgery
9. Planned hospitalization or invasive surgery during the study
10. Severe acute illness unrelated to CDI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zain Kassam, MD, MPH, Study Director — Finch Therapeutics
Locations (54):
- United States (50):
  - Scottsdale, Scottsdale, Arizona
  - Los Angeles, Los Angeles, California
  - Murrieta, Murrieta, California
  - Oakland, Oakland, California
  - San Diego, San Diego, California
  - San Francisco, San Francisco, California
  - Aurora, Aurora, Colorado
  - Bridgeport, Bridgeport, Connecticut
  - Hamden, Hamden, Connecticut
  - Washington DC, Washington D.C., District of Columbia
  - Jacksonville, Jacksonville, Florida
  - Naples, Naples, Florida
  - Pinellas Park, Pinellas Park, Florida
  - Tampa, Tampa, Florida
  - Atlanta, Atlanta, Georgia
  - Idaho Falls, Idaho Falls, Idaho
  - Burr Ridge, Burr Ridge, Illinois
  - Chicago, Chicago, Illinois
  - Evanston, Evanston, Illinois
  - Maywood, Maywood, Illinois
  - Indianapolis, Indianapolis, Indiana
  - West Des Moines, West Des Moines, Iowa
  - Shawnee, Shawnee Mission, Kansas
  - New Orleans, New Orleans, Louisiana
  - Boston, Boston, Massachusetts
  - Detroit, Detroit, Michigan
  - Royal Oak, Royal Oak, Michigan
  - Rochester, Rochester, Minnesota
  - St. Paul, Saint Paul, Minnesota
  - Butte, Butte, Montana
  - Morristown, Morristown, New Jersey
  - Somers Point, Somers Point, New Jersey
  - New York, New York, New York
  - Bronx, The Bronx, New York
  - Chapel Hill, Chapel Hill, North Carolina
  - Kinston, Kinston, North Carolina
  - Pinehurst, Pinehurst, North Carolina
  - Winston-Salem, Winston-Salem, North Carolina
  - Cincinnati, Cincinnati, Ohio
  - Poland, Poland, Ohio
  - Portland, Portland, Oregon
  - Providence, Providence, Rhode Island
  - Nashville, Nashville, Tennessee
  - San Antonio, San Antonio, Texas
  - Ogden, Ogden, Utah
  - Salt Lake City, Salt Lake City, Utah
  - Annandale, Annandale, Virginia
  - Charlottesville, Charlottesville, Virginia
  - Seattle, Seattle, Washington
  - Grafton, Grafton, Wisconsin
- Canada (4):
  - Calgary, Calgary, Alberta
  - Halifax, Halifax, Nova Scotia
  - London, London, Ontario
  - Toronto, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- CP101: Full Spectrum Microbiota Capsule, Full Spectrum Microbiota: Orally administered donor derived microbiota
Period: Week 8
Arm/Group | CP101
Started | 132
Completed | 123
Not Completed | 9
Period: Week 24
Arm/Group | CP101
Started | 123
Completed | 112
Not Completed | 11

BASELINE CHARACTERISTICS:
Population: Modified Intent to Treat (mITT) population
Arm/Group | CP101
Number analyzed (Participants) | 132
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66 (15.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 99
  Male | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 126
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 127
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Canada | 9
  United States | 123
Total number of C. difficile Infection (CDI) episodes in previous 6 months [Count of Participants; unit: Participants]
  1 | 2
  2 | 44
  3 | 49
  >3 | 37

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Absence of Recurrence Through Week 8 Based on Adjudication
Description: Defined in the protocol as sustained clinical cure. Clinical cure means a patient did not experience a recurrence of C. diff during this time period.
Time Frame: Up to Week 8
Population: mITT
Measure: Count of Participants; unit: Participants
Arm/Group | CP101
Number analyzed (Participants) | 132
Participants | 106

2. Primary Outcome: Occurence of Treatment Emergent Adverse Events (TEAEs)
Time Frame: Week 8
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | CP101
Number analyzed (Participants) | 132
Participants | 88

3. Secondary Outcome: Number of Participants With Absence of Recurrence Through Week 24 Based on Adjudication
Description: as for outcome 1
Time Frame: Up to Week 24
Population: mITT
Measure: Count of Participants; unit: Participants
Arm/Group | CP101
Number analyzed (Participants) | 132
Participants | 104

ADVERSE EVENTS:
Time Frame: Up to Week 24
Arm/Group | CP101
All-Cause Mortality (participants affected / at risk) | 1/132
Serious Adverse Events (participants affected / at risk) | 17/132
Other Adverse Events (participants affected / at risk) | 97/132
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CP101 (N=132)
Anaemia (Blood and lymphatic system disorders) | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 2
Acute left ventricular failure (Cardiac disorders) | 1
Angina pectoris (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Atrial flutter (Cardiac disorders) | 1
Bradycardia (Cardiac disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1
Rectal prolapse (Gastrointestinal disorders) | 1
Rectal ulcer (Gastrointestinal disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Clostridium difficile infection (Infections and infestations) | 1
Clostridium difficile colitis (Infections and infestations) | 2
Osteomyelitis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 1
Postoperative fever (Injury, poisoning and procedural complications) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Encephalopathy (Nervous system disorders) | 1
Metabolic encephalopathy (Nervous system disorders) | 1
Suicidal ideation (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Haematoma (Vascular disorders) | 1
Hypertensive emergency (Vascular disorders) | 1
Hypovolaemic shock (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CP101 (N=132)
Diarrhoea (Gastrointestinal disorders) | 52
Abdominal pain (Gastrointestinal disorders) | 43
Defaecation urgency (Gastrointestinal disorders) | 33
Nausea (Gastrointestinal disorders) | 24
Abdominal distension (Gastrointestinal disorders) | 23
Abdominal tenderness (Gastrointestinal disorders) | 17
Anal incontinence (Gastrointestinal disorders) | 13
Vomiting (Gastrointestinal disorders) | 12
Haematochezia (Gastrointestinal disorders) | 10
Urinary tract infection (Infections and infestations) | 7
Decreased appetite (Metabolism and nutrition disorders) | 24
Dehydration (Metabolism and nutrition disorders) | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The disclosure restrictions on the PI are: (i) the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period of up to eighteen months from the lock-down of all study data and (ii) the sponsor can require the removal of its confidential information from results communications and may delay release for a period of up to 60 days for the purpose of filing patent applications.

DOCUMENTS (2):
  • Study Protocol (2019-12-20): https://cdn.clinicaltrials.gov/large-docs/06/NCT03497806/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-05): https://cdn.clinicaltrials.gov/large-docs/06/NCT03497806/SAP_001.pdf